CLINICAL TRIAL: NCT00765336
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Examine the Effects of Minocycline Extended-Release Tablets on Spermatogenesis in Human Males
Brief Title: A Study to Examine the Effects of Minocycline Extended-Release Tablets on Sperm Production in Human Males.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medicis Pharmaceutical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-0104-18; IND 65,398
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2011-12-07 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-11

CONDITIONS: Human Volunteer
Keywords: Spermatogenesis in Healthy Males

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline Extended-Release Tablets (Active Comparator)
  Interventions: Drug: minocycline extended release
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: minocycline extended release — 1 mg/kg extended release minocycline HCL, once daily for 84 days.
  Arms: Minocycline Extended-Release Tablets
Drug: Placebo — placebo comparator for 1 mg/kg extended release minocycline HCL, once daily for 84 days.
  Arms: Placebo

SUMMARY:
Researchers want to find out how Minocycline Extended-Release Tablets affect sperm-production in healthy males.

The study will include Minocycline Extended-Release Tablets, a new once-daily formulation of minocycline, compared with a placebo or inactive pill.

Approximately 170 healthy adult males will be assigned by chance (like flipping a coin) to 2 treatment groups with approximately 85 subjects per group. You will be treated with either Minocycline Extended-Release Tablets or placebo once daily. Screening will occur within 14 days prior to the first dose of study drug.

Required study activities include:

* Written informed consent
* Weight
* Two semen collections within 48-72 hours of one another at the screening visit and Days 84,112, 140, and 168
* Blood draws at the screening visit and Days 84, 112, 140, and 168
* Genital examination (excluding prostate) at screening and at the Day 84 and Day 112 visits
* Medical history

You will continue in the treatment phase of the study for 12 weeks.

You will return to the clinic 4 weeks and 8 weeks after completion of the treatment phase of the study, with the final study visit approximately 12 weeks after the last dose.

Participation will be for 24-weeks.

Up to 10 investigational sites will enroll subjects into the study.

ELIGIBILITY:
Inclusion Criteria:

* Males at least 18 years of age
* Weight 45 kg - 136.36 kg (99-300 lbs)
* Must understand and give consent voluntarily to be in the study and to comply with study requirements
* Subjects must ejaculate between 48 and 72 hours prior to collection of the first specimen (Pre-Collection Ejaculation) and refrain from further ejaculation until Specimen 1 is collected. The second ejaculation sample Specimen 2) must be collected between 48 hours and 72 hours after Specimen 1. No ejaculation is permitted between Specimen 1 and Specimen 2
* Must refrain from using saunas or hot tubs during the duration of the study 168 days)
* Must be a non smoker
* Must be medically healthy as determined by the investigator physician (via medical history and clinical laboratory tests)
* Must have sperm parameters (average of Specimen 1 and Specimen 2) within clinically acceptable limits at screening defined as:
* Total sperm concentration ≥20 x 106/mL10
* % motile ≥50%10
* % normal morphology >4.4%14

Exclusion Criteria:

* Known allergy/sensitivity to minocycline or any of the other drug product components
* Use of antacids or other dietary supplements containing aluminum, calcium, iron, or magnesium
* History of vestibular incidents including vertigo, lightheadedness, nausea, or vomiting within the 30 days prior to enrollment
* Known history of alcohol or drug dependency, significant within the past 2 years
* Known history or current risk of hepatic dysfunction
* Known history or current risk of renal dysfunction, e.g., uncontrolled diabetes
* Systemic lupus erythematosis (SLE) or a positive ANA at screening
* Receipt of any experimental drugs within 120 days prior to Study Day 0
* Non-LFT clinical laboratory values outside the normal range and determined to be of clinical significance
* Liver function tests greater than 1.5 times the upper limit of normal (ALT, AST, GGT)
* Use of tetracyclines, erythromycin within 12 weeks of Day 0

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sanstead, BSN, CCRP, Study Chair — Medicis Pharmaceutical
Locations (10):
- United States (10):
  - West Coast Clinical Research, Tarzana, California
  - University of Minnesota, Minneapolis, Minnesota
  - Women's Health Research Center, LLC, Lawrenceville, New Jersey
  - Weill Cornell Medical College, Great Neck, New York
  - Maze Laboratories, Purchase, New York
  - Tri-State Urologic Services, PSC, Inc., Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Urology San Antonio Research, PA, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Urology of Virginia, PC, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Minocycline Extended-Release Tablets: daily dose of 1 mg/kg minocycline extended-release tablets
- Placebo: daily dose of Placebo
Period: Overall Study
Arm/Group | Minocycline Extended-Release Tablets | Placebo
Started | 91 | 89
Completed | 72 | 73
Not Completed | 19 | 16
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Lost to Follow-up | 7 | 9
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline Extended-Release Tablets | Placebo | Total
Number analyzed (Participants) | 91 | 89 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 89 | 180
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.4 (11.0) | 32.2 (9.0) | 32.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 91 | 89 | 180
Region of Enrollment [Number; unit: participants]
  United States | 91 | 89 | 180

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Screening in Sperm Concentration.
Time Frame: Baseline and 12 Weeks
Population: The enrollment was designed to ensure study completion of approximately 150 subjects. Actual enrollment was 180 subjects (92 in the minocycline group, 88 in the placebo group). A total of 145 subjects (72 in the minocycline group, 73 in the placebo group) comprised the completed population group.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Minocycline Extended-Release Tablets | Placebo
Number analyzed (Participants) | 72 | 73
Percent change | 9.8 (58.3) | -1.3 (47.7)

ADVERSE EVENTS:
Time Frame: Posted adverse event data was collected during the treatment phase (through week 12)
Arm/Group | Minocycline Extended-Release Tablets | Placebo
Serious Adverse Events (participants affected / at risk) | 0/91 | 2/89
Other Adverse Events (participants affected / at risk) | 33/91 | 27/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline Extended-Release Tablets (N=91) | Placebo (N=89)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not related.
Back Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Not Related
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline Extended-Release Tablets (N=91) | Placebo (N=89)
Infections and Infestations (Infections and infestations) | 8 | 9
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 3 | 2
Investigations (Investigations) | 5 | 2
Nervous System Disorders (Nervous system disorders) | 4 | 3
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 11 | 4
Gastrointestinal Disorders (Gastrointestinal disorders) | 8 | 6
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Specific restrictions and agreements are specified in each investigator's contract.